CLINICAL TRIAL: NCT07065877
Title: Clinical and Radiographic Assessment Of Immediate Implant With Topical Vitamin D and Xenograft Mixture: A Randomized Controlled Study
Brief Title: Effect of Vitamin D on Crestal Bone Loss Around Immediate Implant After Mandibular Premolars and Molars Extraction
Acronym: vitD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohamed elsaeed, master candidate oral and maxillofacial surgery, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 961/2025
Record Dates: First submitted 2025-06-27; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Crestal Bone Loss
MeSH Terms: interventions — Transplantation, Heterologous; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: vitamin D solution mixed with xenograft around immediate implant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- vit D mixed with xenograft (Active Comparator): Topical application of vitamin D solution mixed with xenograft in the jumping gap around immediate implant
  Interventions: Drug: vit D mixed with xenograft
- only xenograft without vit D (Placebo Comparator): grafting the jumping gap with xenograft only around immediate implant
  Interventions: Drug: only xenograft without vit D

INTERVENTIONS:
Drug: vit D mixed with xenograft — Topical application of vitamin D solution mixed with xenograft in the jumping gap around immediate implant
  Other Names: cholecalciferol
  Arms: vit D mixed with xenograft
Drug: only xenograft without vit D — grafting the jumping gap with xenograft only around immediate implant
  Other Names: xenotransplant
  Arms: only xenograft without vit D

SUMMARY:
What is the difference between grafting the jumping gap upon using xenograft mixed with topical vitamin D clinically regarding crestal bone level and implant stability, radiographically regarding crestal bone level after implant insertion in the posterior region of mandible?

DETAILED DESCRIPTION:
Effect of Vitamin D on Bone Regeneration .Vitamin D is known for its role in the skeletal system. Vit D deficiency is also widely researched for its effects on the healing of fractures, bone defects and osseointegration of implants. There are studies that investigated the effects of dietary supplementation with vitamin D to reduce vitamin D deficiency but increasing the serum level of this vitamin takes time therefore, an attempt has been made to combat the effect of vitamin D deficiency through topical application. up to the knowledge, upon search of literatures, there is not enough studies that correlate topical application of vitamin D with xenograft mixture as filling space material. this study is to Assess immediate implant with topical vitamin D and xenograft mixture clinically and Radiographically.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologist (ASA) I , II
* Both Genders. 3- Patients having unrestorable tooth on the posterior mandibular region
* Age>20
* The patient who have complete their facial growth and teeth eruption
* No bone disease or lesion in propose implant site

Exclusion Criteria:

* Poor oral hygiene patients and/or patients
* Patients with active acute infection.
* Patients with bad oral habits.
* Pregnant or lactating women.
* Heavy smokers.
* Alcohol and drug addicts.
* Diabetes disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
clinically: A)Loss of crestal bone. B)Stability of implant. Radiographically: crestal bone loss by periapical radiograph in millimeters. | clinically: Loss of crestal bone by periodontal prop assessed in millimeters in six months Stability of implant by OSTTEL assessed as ISQ values in six months crestal bone loss in millimeters will be one ,three months and six months.
  the loss of crestal bone after implant insertion using periodontal probe in millimeters.
  implant stability using OSTELL device. Postoperative follow up using periapical radiographs to evaluate crestal bone loss in millimeters will be after, one ,three months and six months by standardized parallel periapical digital technique radiograph .The radiographs will be done by using: The Kavo Scan eXamTM One and the Rinn extension cone paralleling (XCP)periapical film holder will be used to achieve standardization of digital radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed elsaeed ibrahim, master, Principal Investigator — Suez Canal University
Locations (1):
- oral and maxillofacial surgery depertment of oral and dental medicine faculty Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No